CLINICAL TRIAL: NCT04708912
Title: TUSEB-Nasopharynx Microbiota Component and in Vitro Cytokines Production in Coronavirus Disease (COVID-19)
Brief Title: Nasopharynx Microbiota Component and in Vitro Cytokines Production in Coronavirus Disease (COVID-19)
Acronym: 8796
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Hursitoglu, Associate Professor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 8796
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Microbiota and RNA sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Mild-Moderate COVID-19
  Interventions: Other: Observation
- 2: Severe COVID-19
  Interventions: Other: Observation
- 3: Convalsent (COVID-19)
  Interventions: Other: Observation
- 4: Healthy persons

INTERVENTIONS:
Other: Observation — The study parameters will be obtained at the time of recuirement (Basal)
  Groups: 1; 2; 3

SUMMARY:
The investigators will study nasopharunx microbiota composition, RNA sequences and in vitro cytokines production by peripheral blood cells of COVID-19 patients (both mild-moderate and severe cases) (comparing with convalescent patients and healthy controls).

DETAILED DESCRIPTION:
The investigators will compare study parameters (basal) between mild-moderate and severe COVID-19 patients and with other study groups (i.e. convalescent and healthy controls). Nasopharunx microbiota dysbiosis, in vitro cytokines production profile, and peripheral blood flocytometric results of the four study groups will be compared.

In vitro cytokines production will be studied and compared in Nill (No antigens) and Mitojen (Cocktail of antigens) pre-prepared test tubes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give a written consent

Exclusion Criteria:

* In ability to give a written consent
* Using of medications that affect the results of study parameters
* Presence of malignancy or tuberculosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (18-80 yerars ), both gender
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Determination of peripheral blood RNA microarray assay | First day
  Four study groups, microarray Analysis .
Determination of nasopharunx Microbiota analysis | 1st day
  Four study groups, metagenomic analysis, to determine abundance and decrease of some species.
Determination of in vitro cytokines production | First day
  IL-2, IL-7, IL-10, granulocyte-colony stimulating factor, interferon-p inducible protein 10, monocyte chemo-attracting protein 1, macrophage inflammatory protein 1-α and tumor necrosis factor-α in Nill (no angijen) and Mitojen (Cocktails of antigens)tubes (between 4 study groups)
Determination of peripheral blood cytometry | First day
  Four study groups, peripheral blood cytometry; CD3, CD4, CD8, and CD45 rates.
Relation between study parameters | First day parameters
  determining the realtion between microbiotme dysbiosis, in vitro cytokines production and peripheral leymphocytes (CD3,CD4, CD8, and CD45) rates and the severity of COVID-19( if any)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Hursitoglu, MD, Principal Investigator — Basaksehir Cam and sakura Sehir Hospital
Locations (1):
- Bakirkoy Dr.sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Microbiota and viral infections